CLINICAL TRIAL: NCT05278936
Title: A Simplified Sclerocorneal Incision/Tunnel in Performing Congenital/Pediatric Cataract Surgery
Brief Title: New Technique in Congenital/Pediatric Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omer Othman Abdullah (Other)
Responsible Party: Sponsor-Investigator, Omer Othman Abdullah, Associate consultant ophthalmologist, Ibinsina Modern Eye and Retina Center
Organization: Ibinsina Modern Eye and Retina Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMER 1
Record Dates: First submitted 2022-02-23; First posted 2022-03-14 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Pediatric Cataract; Congenital Cataract
Keywords: Corneoscleral incision; Cataract surgery; Vitreorrhexis; Anterior vitrectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A simplified sclero-cornel tunnel/incision in performing the congenital/pediatric cataract surgery (Other): Participitant
  Interventions: Other: The cataract surgery and the anterior vitrectomy

INTERVENTIONS:
Other: The cataract surgery and the anterior vitrectomy — Surgical

SUMMARY:
In pediatric/congenital cataract surgery; multiple surgical interventions are performed, which needs multiple general anesthesias. Here, we describe a new technique, to end the operation in one session.

DETAILED DESCRIPTION:
Generally, in congenital/pediatric cataract surgery, it might be possible to different multiple procedures with multiple general anesthesias. Here, the investigators found a new procedure to perform the cataract removal, intraocular implantation, and the anterior vitrectomy all in one session through a sclero-corneal tunnel. The corneoscleral tunnels are covered by the conjunctiva to abolish the need for both suturing and repeated general anesthesia to remove corneal sutures.

ELIGIBILITY:
Inclusion Criteria:

* Congenital/pediatric cataract

Exclusion Criteria:

* Aphakic and pseudophakic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-10-01 (Actual)

PRIMARY OUTCOMES:
Slit-lamp examination | The fourth weeks postoperatively
  To check the intra-ocular lens positioning

CONTACTS AND LOCATIONS:
Overall Officials: Omer Abdullah, M.Sc., Principal Investigator — Ibinsina Modern Eye and Retina Center; Huseyin Oksuz, MD, Study Director — Dunya Goz Hospital
Locations (1):
- Ibinsina Modern eye and retina center, Erbil, Iraq

IPD SHARING:
Plan to Share IPD: No